CLINICAL TRIAL: NCT05031793
Title: Establishing the Collaborative Care Model of TCM and Western Medicine for Pediatric Allergic Rhinitis With Sleep Disorder
Brief Title: Establishing the Collaborative Care Model for Pediatric Allergic Rhinitis With Sleep Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Rong Yen, Attending physician, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH106-REC2-140
Record Dates: First submitted 2018-05-16; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis; Sleep Disorder
Keywords: Allergic rhinitis; Sleep disorder; Obstructive sleep apnea; Integrative care clinic; TCM; Western medicine
MeSH Terms: conditions — Rhinitis, Allergic; Sleep Wake Disorders; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care of TCM and Western Medicine (Experimental)
  Interventions: Other: TCM; Other: Western medicine
- Western medicine (Active Comparator)
  Interventions: Other: Western medicine

INTERVENTIONS:
Other: TCM — TCM include oral chinese herb, laser acupuncture, tuina, nasal steam inhalation.
  Arms: Collaborative Care of TCM and Western Medicine
Other: Western medicine — Western medicine include nasal spray steroid, oral antihistamine

SUMMARY:
The purpose of study is to compared the impact of the integrative care clinic to ordinary western medicine among patients of moderate persistent allergic rhinitis combined with sleep disorder and establishing the collaborative care model of TCM and western medicine for pediatric allergic rhinitis with sleep disorder.

Investigators invited children aged below 18 years old to the integrative care clinic as experimental group, who have persistent moderate allergic rhinitis, more than 60 scores of the OSA-18 sleep questionnaire, and can accept integrative therapy. The controlled group is patients who receive ordinary western treatment. Investigators compare these two groups by questionnaires of OSA-18,SN-5, PADQLQ,SNAP-IV, the dose of nasal corticosteroid , and polysomnography.

DETAILED DESCRIPTION:
In Taiwan, there are many patients suffer from pediatric allergic rhinitis and lead to the medical heavy budget. The persistent symptoms would cause sleep disorder or complicated with pediatric obstructive sleep apnea. It would affect the growth development ,attention deficiency, or psychiatric cognition problems. Obstructive sleep apnea for a long time would result in cardiovascular, endocrine, and metabolic complications if not well-treated.

Patients of allergic rhinitis combined with sleep disorder are classified to moderate persistent type by ARIA, who are intractable to ordinary treatment. Investigators invited them to the integrative care clinic. In addition to the ordinary western medicine, the therapies in the integrative care clinic included herbal medicine, nasal aerosol inhalation, acupuncture, and health care education. The purpose of our study is to compared the impact of the integrative care clinic to ordinary western medicine among patients of moderate persistent allergic rhinitis combined with sleep disorder and establishing the collaborative care model of TCM and western medicine for pediatric allergic rhinitis with sleep disorder.

Investigators invited children aged below 18 years old to the integrative care clinic as experimental group, who have persistent moderate allergic rhinitis, more than 60 scores of the OSA-18 sleep questionnaire, and can accept integrative therapy. The controlled group is patients who receive ordinary western treatment. Investigators compare these two groups by questionnaires of OSA-18,SN-5, PADQLQ,SNAP-IV, the dose of nasal corticosteroid , and polysomnography.

Investigators hoped to prove the effect of integrative care clinic and to upgrade the quality and efficacy of the treatment among persistent moderate allergic rhinitis children.

ELIGIBILITY:
Inclusion Criteria:

1. age <18 years old
2. ARIA (2014) diagnostic criteria belong to moderate, persistent
3. OSA-18 score ≥60

Exclusion Criteria:

1. cranial-facial anomaly
2. secondary obstruction sleep apnea due to muscle weakness of upper airway, such as Down syndrome or cerebral palsy
3. psychiatric disease or behavior disorder
4. allergy to TCM or ordinary western medicine treatment
5. asthma

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
The change of SN-5 scores | week 8
  SN-5 questionnaire is a tool to evaluate quality of life of sinus and nasal symptoms

SECONDARY OUTCOMES:
The change of scores of Pediatric allergic disease quality of life questionnaire (PADQLQ) | week 8
  Pediatric allergic disease quality of life questionnaire (PADQLQ) is a validated tool to evaluate quality of life of pediatric allergic disease.
The change of scores of questionnaire of pediatric obstructive sleep apnea (OSA-18) | week 8
  Obstructive Sleep Apnea-18
The change of scores of Pediatric Sleep Questionnaire | week 8
  Pediatric Sleep Questionnaire is a validated questionnaire to evaluate sleep quality among children
The change of hyperactivity-inattentive condition | week 8
  SNAP-IV is a validated tool designed by Swanson, Nolan and Pelham ,is the questionnaire used to evaluate hyperactivity-inattentive condition .
dosage of intra-nasal corticosteroid | week 8
  Weight change of intra-nasal corticosteroid before and after study
Apnea-Hyponea index | week 12
  Apnea-Hyponea index is evaluated by polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Rong Yen, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan